CLINICAL TRIAL: NCT01793896
Title: Mitochondrial Biogenesis, Reduction of Muscle Oxidative Damage and Improvement in Adipose Tissue Functional Profile, Account for the Beneficial Effects of Exercise and Healthy Diets
Brief Title: Beneficial Effects of Exercise and Healthy Diets on Muscle and Adipose Tissue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Serious difficulties for patient recruitment
  to recruit patients
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, MARIA PIA DE LA MAZA, Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Fondecyt 1130284; INSTITUTE OF NUTRITION 2013 (Other: INTA)
Record Dates: First submitted 2013-02-11; First posted 2013-02-18 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Ageing; Mitochondrial density; Oxidative damage; Inflammatory mediators; AMPK; Adipogenesis
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Mediterranean; Diet; Exercise

STUDY DESIGN:
Intervention Model Description: After a placebo phase with no intervention in the first 25 subjects recruited, overweight or obese patients were randomly assigned to one of 3 treatments: hypocaloric diet, high intensity interval training or both interventions simultaneously, for 3 months.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control period (Sham Comparator): control period with no intervention. Comparison of parameters at entrance and one month later without any intervention
  Interventions: Behavioral: Control period
- Diet group (Experimental): Mediterranean diet prescription during 3 months
  Interventions: Behavioral: Diet Group
- Exercise group (Experimental): Subjects will be trained 3 times a week during 3 months
  Interventions: Behavioral: Exercise group
- Diet + Exercise (Experimental): Both a dietary prescription plus exercise training during 3 months
  Interventions: Behavioral: Diet + Exercise

INTERVENTIONS:
Behavioral: Control period — Analysis at recruitment and after a month without any intervention
  Other Names: Before randomization
  Arms: control period
Behavioral: Diet Group — selected subjects will adopt a Mediterranean low-AGE diet. We will not include red wine in the Mediterranean diet (7 Kilocalories (KCal)/g), in order to attain more weight loss. Each subject will be instructed to reduce 500 Kcal of their estimated total daily energy requirements, so theoretically they will be able to reduce 5 - 10 % of their body weight in 3 months.
  Other Names: Mediterranean diet
  Arms: Diet group
Behavioral: Exercise group — The intervention will consist of 3 weekly 1 hour sessions (5 minutes of preconditioning, followed by 20 minutes cycling, brisk walking or jogging at 65-70 % maximal aerobic capacity, then 25 minutes resistance weight-lifting exercises and finally 10 minutes of stretching). Exercise intensity will be increased weekly according to the Borg Scale intensity. The exercise intervention will be supervised by physical education teachers, registering attendance at every session.
  Arms: Exercise group
Behavioral: Diet + Exercise — these patients will be incorporated to receive both Mediterranean diet plus exercise interventions
  Arms: Diet + Exercise

SUMMARY:
Both dietary caloric restriction (CR) and physical exercise (PE) exert beneficial effects, which retard or prevent age-related diseases and prolong life span. Subjects with the metabolic syndrome age prematurely, therefore preventive measures should be initiated early. The present study intends to demonstrate that physical exercise and/or Mediterranean diet, in middle aged volunteers with the metabolic syndrome, preserve adequate adipose tissue functionality and retard skeletal muscle aging (assessed by mitochondrial biogenesis and accumulation of ROS), by activating several pathways, homologous to CR. The investigators plan to study this by using two approaches: 1) A cross- sectional model, in which the expression of the mentioned metabolic mediators, indicators of muscle mitochondrial biogenesis and muscle oxidative damage will be compared between men with different body compositions, fat distribution, muscle strength and exercise capacity (VO2max). Also, in these men the investigators will assess the expression of uncoupling protein 1 (UCP1) in subcutaneous white adipose tissue (as a measure of adaptive thermogenesis), and inflammatory markers (Interleukin 1-6, Interleukin 1ß and CCL2 chemokine (C-C motif ligand 2)) in preperitoneal adipose tissue, plus inflammation and adipogenesis potential of their cultured preadipocytes. Moreover, in vitro studies will evaluate the functional effects of exposure of a cell lyne of human adipocyte cells (LS14)to factors secreted by media conditioned by the patients´ adipose tissue explants. 2) A prospective intervention in overweight/moderately obese middle aged volunteers that will be assigned to a weight-maintenance period (as a control group), and then randomly y assigned to a Mediterranean diet, exercise training or diet plus training. Before and after 3 months of intervention the investigators will obtain muscle tissue samples to study the expression of Peroxisome proliferator activated receptor (PPAR) gamma coactivator 1 alpha (PGC1), uncoupling protein 3 (UCP3), AMP activated protein kinase (AMPK), Sirtuin 1 (SIRT-1), mitochondrial DNA and oxidative damage indicators (8-oxo-7,8-dihydro-2-deoxyguanosine (oxodG), carboxymethyllysine (CML and its receptor (RAGE)). In vitro studies will evaluate the effect of circulating factors from the patients (serum) on LS14 inflammatory and adipogenic potential, at baseline and after 3 months of intervention.

DETAILED DESCRIPTION:
METHODOLOGY:

This study will be composed of 2 parts:

I - CROSS SECTIONAL STUDY The aim of this section is to compare men with different body compositions, fat distribution and exercise capacity with respect to their muscle mitochondrial biogenesis, oxidative damage and energy flux regulator molecules, together with their adipose tissue inflammation, adipokine expression and thermogenic potential.

Inclusion criteria :

* male sex
* age 25 - 50 years
* BMI from 20 - 35 kg/mt2
* indication for surgery of an inguinal hernia

Exclusion criteria:

* diabetes mellitus
* chronic neuromuscular or neurological deficits precluding normal physical activity
* heavy smoking (> 5 cigarettes per day)
* alcohol intake > 30 g/day
* chronic diseases such as cancer, HIV-AIDS, renal, pulmonary, cardiac or hepatic conditions.

Before the operation and after signing a written informed consent, the following assessment will be performed:

1. Medical history including medication intake and complete physical examination.
2. Dietary recall of habitual intake and calculation of AGEs ingestion.
3. Regular physical activity assessment using the International Physical Activity Questionnaire
4. Anthropometrics (height, weight, waist circumference)
5. Fasting blood sampling for routine determinations (haemoglobin,lipoproteins, creatinine,prothrombin, TSH), AGEs concentrations (CML) free fatty acids, adiponectin and 8- Isoprostanes.
6. Fasting and post glucose serum sampling for glucose and insulin measurements, and calculation of Homeostasis Model Assessment (HOMA-IR) and the Matsuda Index for determination of peripheral insulin sensitivity.
7. Resting and exercise indirect calorimetry for estimation of resting energy expenditure, respiratory quotient and VO2 max.
8. Handgrip and quadriceps muscle strength
9. Dual X-Ray Energy Densitometry (DEXA) for estimation of body composition
10. CT scan of abdominal region at L4 level for measurement of visceral and subcutaneous fat areas and estimation of liver fat infiltration.
11. Ultrasound intensity analysis in thigh ultrasonography indicating muscle fat infiltration. After the initial evaluation, subjects will be classified as with or without the metabolic syndrome, according to the international guidelines guidelines, for further analysis of data.

A few days later, during the surgical procedure, a sample of muscle tissue (approximately 200 mg of internal abdominal oblique) will be obtained for measurement of:

1. Fiber type
2. Messenger Ribonucleic acid (mRNA) expression of PGC-1-alpha, SIRT-1, UCP-3 and AMPK
3. Mitochondrial density by measurement of mitDNA and Cytochrome C activity
4. Oxidative damage (8-oxodG, CML and RAGE).

During the same operation, 2 samples of adipose tissue will also be obtained, one subcutaneous (at the site of the incision) and the other preperitoneal (at the inguinal sac), for in vitro studies:

1. UCP1 and inflammatory marker (interleukin 6, 1ß, CCL2) expression in mature adipocytes
2. Inflammatory profile and adipogenic potential (expression of lipoprotein lipase, PPAR gamma and adiponectin) in cultured preadipocytes
3. Adipogenic potential and inflammatory expression profile of LS14 adipose cells exposed to conditioned media from adipose tissue explants.

A small part of these adipose tissue samples will be placed in formaldehyde, fixed and stained with H.E for histologic estimation of adipocyte cell size.

II - INTERVENTION STUDY This section intends to demonstrate the effects of a low-AGEs Mediterranean diet and/or exercise, over skeletal muscle metabolic profile and adipogenic/inflammatory features of adipocytes.

Inclusion criteria:

* Overweight or obese men and women
* Ages 25 - 50 years
* Interest in losing weight

Exclusion criteria:

* weight fluctuations (> 3 k in the last 3 months)
* diabetes mellitus
* chronic neuromuscular or neurologic diseases
* heavy smoking (> 5 cigarettes per day)
* alcohol intake > 30 g/day
* chronic diseases such as cancer, HIV, renal, pulmonary, cardiac or hepatic conditions.

Subjects will be invited to participate in a trial using a Mediterranean low-AGEs diet and/or physical exercise during 3 months. After signing a written informed consent,subjects will be allocated to one of these interventions, which will be randomly selected, and the following assessment will be performed, at baseline and after 3 months of intervention:

1. Medical and medication intake history and complete physical examination.
2. Dietary recall of habitual intake and calculation of AGEs ingestion.
3. Physical activity questionnaire (IPAQ)
4. Anthropometrics (height, weight, waist circumference)
5. Fasting blood sampling for routine determinations (haemoglobin, lipoproteins, creatinine, prothrombin and TSH), AGEs concentrations (CML), free fatty acids, adiponectin, 8-Isoprostanes and serum for in vitro adipose tissue studies (see below).
6. Fasting and post glucose blood sampling for glucose and insulin measurements, and calculation of HOMA-IR and the Matsuda Index for determination of peripheral insulin sensitivity.
7. Dual X-Ray Energy Densitometry (DEXA) for estimation of body composition
8. CT scan of abdominal region at L4 level for measurement of visceral and subcutaneous fat areas and estimation of liver fat infiltration
9. Resting and exercise indirect calorimetry for estimation of resting energy expenditure, respiratory quotient and VO2 max.
10. Handgrip and quadriceps muscle strength
11. Ultrasound intensity analysis in thigh indicating muscle fat infiltration
12. Ultrasound guided quadriceps muscle biopsy to measure mitochondrial density (mitDNA) and expression of PGC-1

ELIGIBILITY:
Inclusion Criteria:

CROSS SECTIONAL: male sex, age 25 -50 years, with BMI ranging from 20 to 35 kg/mt2. INTERVENTION STUDY: Overweight or obese men and women aged 25 - 50 years interested in losing weight,will

Exclusion Criteria:

CROSS SECTIONAL : diabetes mellitus, chronic neuromuscular or neurological deficits precluding normal physical activity, heavy smoking (> 5 cigarettes per day), alcohol intake > 30 g/day and chronic diseases such as cancer, HIV-AIDS, renal, pulmonary, cardiac or hepatic conditions.

INTERVENTION STUDY: weight fluctuations (> 3 k in the last 3 months), diabetes mellitus, chronic neuromuscular or neurologic diseases, heavy smoking (> 5 cigarettes per day) and alcohol intake > 30 g/day, and chronic diseases such as cancer, HIV, renal, pulmonary, cardiac or hepatic conditions.

-

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in mitochondrial density in muscle tissue | 3 months
  As described in the methodology section

SECONDARY OUTCOMES:
Change in Oxidative damage in muscle tissue | 3 months
  As described in the methodology section

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pia de la Maza, Professor, Principal Investigator — University of Chile
Locations (1):
- Institute of Nutrition & Food Technology (INTA), Santiago, Metropolitan Region, Chile